CLINICAL TRIAL: NCT06196307
Title: A Prospective Study of Acute Nontraumatic Chest Pain - Warning and Classification
Brief Title: Early Warning and Classification Model for Acute Non-traumatic Chest Pain
Status: Recruiting | Type: Observational
Sponsor: Xiao-nan He (Other)
Responsible Party: Sponsor-Investigator, Xiao-nan He, Chief physician of Emergency and Critical Care Center of Beijing Anzhen Hospital, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Other Study IDs: F0213-62272327
Record Dates: First submitted 2023-10-27; First posted 2024-01-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain | interventions — Laboratories; Dosage Forms; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- No cardiovascular adverse and cerebrovascular events (MACCE) occurred during the 1-month period: No cardiovascular and cerebrovascular adverse events (MACCE)，which included cardiovascular death, all-cause mortality, nonfatal myocardial infarction, refractory angina, new onset heart failure and stroke. Follow-up visits are conducted by in-person or telephone and registration is carried out.
  Interventions: Combination Product: Clinical evaluation, laboratory and cardiac imaging results, medication, surgery, and any hospitalization
- Group of major cardiovascular and cerebrovascular adverse events (MACCE) occurring during 1 month: Cardiovascular and cerebrovascular adverse events occur, the rest of the same as in the previous group
  Interventions: Combination Product: Clinical evaluation, laboratory and cardiac imaging results, medication, surgery, and any hospitalization

INTERVENTIONS:
Combination Product: Clinical evaluation, laboratory and cardiac imaging results, medication, surgery, and any hospitalization — Examination： Electrocardiogram、 imaging examination、 X-ray, CTA, bedside echocardiography. Laboratory test results of patients, including complete blood count, D-dimer, myocardial injury markers, sST2, MPO, and other indicators. History of cardiovascular and pulmonary vascular drug therapy: Antithrombotic therapy (type, measurement) , Anticoagulation therapy (type, metering), Other drug treatments (type, measurement)

SUMMARY:
Acute non-traumatic chest pain is one of the common causes of presentation in emergency patients, but the causes of acute non-traumatic chest pain are complex, the severity of the condition varies greatly, and the specificity of symptoms is not high. Machine learning and intelligent auxiliary models can greatly shorten the time of clinical decision-making, and improve the accuracy of etiological diagnosis in patients with chest pain, reduce the rate of misdiagnosis and missed diagnosis, and provide a clear direction for further treatment.

DETAILED DESCRIPTION:
Prospective observational studies used outpatient and follow-up information to construct an auxiliary early warning model of acute non-traumatic chest pain based on federated learning, and optimized the accuracy of early warning models through retrospective and prospective studies of large cohort data, and established an efficient and stable early warning and classification model for acute non-traumatic chest pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Symptom onset or worsening within 24 hours before presentation, with a chief complaint of acute chest pain meeting the broad definition of chest pain (2021 AHA)
3. Presentation to the emergency department, with a clinical diagnosis consistent with non-traumatic chest pain
4. Signed informed consent

Exclusion Criteria:

1. traumatic chest pain
2. systemic pain caused by malignant tumors or rheumatic diseases involving the chest
3. Patients were lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population included patients admitted to the chest pain center of the pilot hospital from August 2022 to December 2027 with chest pain (including tingling, burning pain, pressure, tightness, heartburn and similar discomfort) as the main manifestations. Screening of patients with chest pain is intended from the following sources:
  1. outpatients with chest pain;
  2. outpatients with a history of cardiovascular disease;
  3. patients from other departments of the hospital referred to the cardiology outpatient clinic due to acute chest pain.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 30 days after presenting to the emergency departments(ED)
  The primary outcome was a composite of adjudicated major adverse cardiovascular and cerebrovascular events (MACCE), which included cardiovascular death, all-cause mortality, nonfatal myocardial infarction, refractory angina, new onset heart failure and stroke.

OTHER OUTCOMES:
Differences in accuracy in diagnosing acute non-traumatic chest pain using machine learning and intelligence-assisted models and existing scoring systems. | Week 12
  Cross-disciplinary testing

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaonan He, Beijing, Chaoyang, China

IPD SHARING:
Plan to Share IPD: No